CLINICAL TRIAL: NCT02624024
Title: AQT90 FLEX TnI and TnT - Clinical Sensitivity and Specificity Study
Brief Title: Clinical Performance Evaluation of AQT90 FLEX TnI and TnT
Status: Completed | Type: Observational
Sponsor: Radiometer Medical ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: DC-059975
Record Dates: First submitted 2015-12-04; First posted 2015-12-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frozen plasma samples are retained for this study and possible future studies.

GROUPS / COHORTS (1):
- Acute chest pain or equivalent ischemic symptoms: acute chest pain or equivalent ischemic symptoms suggestive of acute coronary syndromes (ACS) or acute myocardial infarction (MI)

SUMMARY:
The AQT90 FLEX Troponin I (TnI) and Troponin T (TnT) Tests are in vitro diagnostic assays intended as an aid in the diagnosis of myocardial infarction (MI) in point-of-care and laboratory settings. The purpose of the study is to establish the clinical performance of the AQT90 FLEX TnI and TnT assays for both whole blood and plasma in the intended use population.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 21 years of age or older.
* Subject is able to understand information given, and willing and able to voluntarily give their consent to participate in this study.
* Subject is presenting to the ED with acute chest pain or equivalent ischemic symptoms suggestive of ACS or MI (e.g., acute chest pain/pressure, shortness of breath, discomfort in upper extremity, jaw or epigastrium, diaphoresis, nausea, vomiting, lightheadedness, dizziness, weakness, and/or syncope).

Exclusion Criteria:

* Subject is pregnant or may be pregnant.
* Subject has an invalid written informed consent or has withdrawn consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 21 years of age or older presenting to the emergency department (ED) with acute chest pain or equivalent ischemic symptoms suggestive of acute coronary syndromes (ACS) or acute myocardial infarction (MI).
Sampling Method: Probability Sample
Enrollment: 1743 (Actual)
Dates: Start 2016-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Diagnosis of acute myocardial infarction (MI) | during the first 24 hours after presentation to the emergency department
  Diagnosis of acute myocardial infarction (MI) that a subject was experiencing at the time of the subject's presentation to the ED, as determined by independent adjudication panel and based on the Third Universal Definition of Myocardial Infarction.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Honor Health Scottsdale Osborn Medical Center, Scottsdale, Arizona
  - Honor Health Scottsdale Shea Medical Center, Scottsdale, Arizona
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indiana University Health Ball Memorial Hospital, Muncie, Indiana
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Cincinnati Department of Emergency Medicine, Cincinnati, Ohio
  - Catholic Health Initiatives Institute for Research and Innovation -CHI Franciscan Health, Tacoma, Washington